CLINICAL TRIAL: NCT00003471
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Adult Patients With Low Grade Astrocytoma
Brief Title: Antineoplaston Therapy in Treating Patients With Low-Grade Astrocytoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066508; BC-BT-16 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Low-Grade Astrocytoma, Nos
Keywords: Recurrent/progressive adult low grade astrocytoma
MeSH Terms: conditions — Astrocytoma; Recurrence | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Adults with a recurrent/progressive low grade astrocytoma will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for adult recurrent/progressive low grade astrocytoma provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of adult recurrent/progressive low grade astrocytoma.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on adults with a recurrent/progressive low grade astrocytoma.

DETAILED DESCRIPTION:
OVERVIEW: This is a single arm, open-label study in which adults with a recurrent/progressive low grade astrocytoma receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in adults with a recurrent/progressive low grade astrocytoma, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in adults with a recurrent/progressive low grade astrocytoma.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed low-grade astrocytoma that has progressed, recurred, or persisted after initial therapy, including radiotherapy
* Previously treated with at least 1 prior standard therapy (e.g., radiotherapy, chemotherapy, immunotherapy, or cytodifferentiating agent)
* Measurable tumor by MRI scan performed within two weeks prior to study entry
* Tumor must be at least 5 mm
* No brain stem tumors

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No renal insufficiency
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No uncontrolled hypertension
* No chronic heart failure
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease (e.g., chronic obstructive pulmonary disease)

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No other concurrent serious disease
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulating agents

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent antineoplastic agents

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* See Disease Characteristics
* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Must recover from prior surgery

Other:

* No prior antineoplastons

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 1996-03; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven patients were recruited between March 1996 and June 2003. All study subjects were seen at the Burzynski Clinic in Houston TX
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Adults with a recurrent/progressive low grade astrocytoma will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 7
Completed | 3
Not Completed | 4
Not completed — Not evaluable | 4

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: Years] | 43.1 [35.2 to 51.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 3
Participants
  Stable Disease | 2
  Progressive Disease | 1

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 7
Percentage of participants
  6 months overall survival | 71.4
  12 months overall survival | 57.1
  24 months overall survival | 42.9
  36 months overall survival | 42.9
  48 months overall survival | 28.6
  60 months overall survival | 28.6

ADVERSE EVENTS:
Time Frame: 7 years, 4 months
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 5/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=7)
Central Venous Catheter: Non-functional (General disorders) | 1 — The Central Venous Catheter: Non-functional was not related to Antineoplaston Therapy.
Central Venous Catheter: Thrombosis/embolism (General disorders) | 1 — The Central Venous Catheter: Thrombosis/embolism was not related to Antineoplaston Therapy.
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 — The Fatigue (asthenia, lethargy, malaise) was not related to Antineoplaston Therapy
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 1 — The Infection (documented clinically): Lung (pneumonia) was not Related to Antineoplaston Therapy.
Hypernatremia (Investigations) | 2 — One of the Hypernatremias was related to Antineoplaston Therapy. One of the Hypernatremias was not related to Antineoplaston Therapy.
Seizure (Nervous system disorders) | 1 — The Seizure was not related to Antineoplaston Therapy.
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 — The Somnolence/depressed level of consciousness was not related to Antineoplaston Therapy.
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 — The Pleural effusion (non-malignant) was not related to Antineoplaston Therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=7)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Hypertension (Cardiac disorders) | 1
Central Venous Catheter: Non-functional (General disorders) | 3
Central Venous Catheter: Thrombosis/embolism (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3
Insomnia (General disorders) | 1
Edema/Fluid retention (General disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 1
Infection (documented clinically): Skin (cellulitis) (Infections and infestations) | 1
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 1
Infection (documented clinically): Urinary tract NOS (Infections and infestations) | 1
Opportunistic infection (Infections and infestations) | 2
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 1
Hypercholesteremia (Investigations) | 1
Hyperglycemia (Investigations) | 3
Hypernatremia (Investigations) | 2
Hypertriglyceridemia (Investigations) | 1
Hypocalcemia (Investigations) | 1
Hypoglycemia (Investigations) | 2
Hypokalemia (Investigations) | 6
Hypophosphatemia (Investigations) | 1
Proteinuria (Investigations) | 1
SGOT (Investigations) | 1
SGPT (Investigations) | 1
Confusion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Mood alteration (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 3
Somnolence/depressed level of consciousness (Nervous system disorders) | 3
Speech impairment (Nervous system disorders) | 1
Vision-blurred vision (Eye disorders) | 1
Pain: Back (Musculoskeletal and connective tissue disorders) | 1
Pain: Chest wall (Musculoskeletal and connective tissue disorders) | 1
Pain: Head/headache (Nervous system disorders) | 2
Pain: Neck (Musculoskeletal and connective tissue disorders) | 1
Pain: Pleura (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Incontinence, urinary (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1
Flu-like syndrome (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No